CLINICAL TRIAL: NCT00561925
Title: A Randomised, Double Blind, Double Dummy, Parallel Group, Active Controlled Trial to Evaluate the Antiviral Efficacy of 400 mg QD neVirapine Extended Release Formulation in Comparison to 200 mg BID neVirapinE Immediate Release in Combination With Truvada® in Antiretroviral Therapy naïve HIV-1 Infected Patients (VERxVE)
Brief Title: VERxVE Study on Efficacy and Safety of Nevirapine XR in Comparison to Nevirapine IR With Truvada in Naive HIV+ Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1100.1486; 2007-003654-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (2):
- nevirapine XR (Experimental): 400 mg QD
  Interventions: Drug: nevirapine XR
- nevirapine IR (Active Comparator): 200 mg BID
  Interventions: Drug: nevirapine IR

INTERVENTIONS:
Drug: nevirapine IR — 200 mg BID
  Arms: nevirapine IR
Drug: nevirapine XR — 400 mg QD
  Arms: nevirapine XR

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 400 mg QD nevirapine extended release (NVP XR) formulation versus 200 mg BID nevirapine immediate release (NVP IR) in ARV therapy naïve HIV-1 infected patients after 48 weeks of treatment. Secondary objectives are to evaluate safety and pharmacokinetics of NVP XR and NVP IR.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent in accordance with Good Clinical Practice and local regulatory requirements prior to trial participation
2. HIV-1 infected males or females >= 18 years of age with positive serology (ELISA) confirmed by Western blot
3. No previous antiretroviral treatment
4. Males with CD4+ counts >50 - <400 cells/ml or females with CD4+ counts >50-<250 cells/ml
5. Adequate renal function defined as a calculated creatinine clearance (CLCr) greater than or equal to 50 mL/min according to the Cockcroft-Gault formula as follows:

   Male: (140 - age in years) x (weight in kg) divided by 72 x (serum creatinine in mg/dl) = CLCr (mL/min).

   Female: (140 - age in years) x (weight in kg) divided by 72 x (serum creatinine in mg/dl) x 0.85 = CLCr (mL/min).
6. Karnofsky score >70 (see Appendix 10.4)
7. An HIV-1 viral load of 1,000 copies/mL
8. Willingness to initiate CD4+ cell count-guided chemoprophylaxis to prevent important opportunistic infections as defined in Appendix 10.2
9. Willingness to abstain from ingesting substances which may alter plasma study drug levels by interaction with the cytochrome P450 system (listed in Appendix 10.3) during the study.
10. For centers participating in the PK substudy only: Written informed consent in accordance with GCP and local legislation for participation in the PK substudy. Refusal to participate in the PK substudy is not an exclusion criterion for participation in the trial. Only study centers with previous experience and equipped in handling PK samples are eligible for participation in the substudy.

Exclusion criteria:

1. Active drug abuse or chronic alcoholism at the investigator's discretion
2. Active hepatitis B or C disease, defined as HBsAg-positive and HBV-DNA-positive or HCV-RNA-positive
3. Female patients of child-bearing potential who: are pregnant at screening; are breast feeding; are planning to become pregnant; are not willing to use a barrier method of contraception, or; are not willing to use methods of contraception other than ethinyl estradiol containing oral contraceptives Note: During participation in this study, females and males have to use barrier methods of contraception in addition or instead of ethinyl estradiol containing oral contraceptives.
4. Laboratory parameters >DAIDS Grade 2
5. ALT/AST > DAIDS Grade 1
6. Hypersensitivity to any ingredients of the test products
7. Previous use of Viramune® (nevirapine) or any other antiretroviral agents (does not include use of single dose NVP for the prevention of mother to child transmission)
8. Resistance to NNRTIs or either one of the components of Truvada® (emtricitabine or tenofovir disoproxil fumarate) or lamivudine (3TC) based on HIV-1 genotypic resistance testing report obtained at screening
9. Patients who are receiving other concomitant treatments which are not permitted, as described in the prescribing information
10. Use of investigational medications (any experimental agent other than the study regimen) within 30 days before study entry or during the trial
11. Use of immunomodulatory drugs within 30 days before study entry or during the trial (e.g., interferon, cyclosporin, hydroxyurea, interleukin 2)
12. Patients who have been diagnosed with malignant disease
13. Patients who in the opinion of the investigator are not candidates for inclusion in the study
14. Patient with Progressive Multifocal Leukoencephalopathy (PML), Visceral Kaposi's Sarcoma (KS), and/or any lymphoma
15. Any AIDS defining illness that is unresolved, symptomatic or not stable on treatment for at least 12 weeks at screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1068 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (202):
- United States (41):
  - 1100.1486.0040 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1100.1486.0013 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1100.1486.0017 Boehringer Ingelheim Investigational Site, Bakersfield, California
  - 1100.1486.0001 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1100.1486.0057 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1100.1486.0059 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1100.1486.0035 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1100.1486.0025 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1100.1486.0034 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1100.1486.0041 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1100.1486.0032 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1100.1486.0028 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1100.1486.0023 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1486.0029 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1486.0048 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1486.0037 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1100.1486.0043 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1100.1486.0012 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1100.1486.0007 Boehringer Ingelheim Investigational Site, Miami Beach, Florida
  - 1100.1486.0039 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1100.1486.0050 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1100.1486.0014 Boehringer Ingelheim Investigational Site, Wilton Manors, Florida
  - 1100.1486.0031 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1100.1486.0010 Boehringer Ingelheim Investigational Site, Macon, Georgia
  - 1100.1486.0053 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 1100.1486.0002 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1100.1486.0026 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1100.1486.0020 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1100.1486.0019 Boehringer Ingelheim Investigational Site, Berkley, Michigan
  - 1100.1486.0006 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1100.1486.0027 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1100.1486.0055 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1100.1486.0003 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 1100.1486.0005 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1100.1486.0004 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1100.1486.0018 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1100.1486.0038 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1100.1486.0044 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1100.1486.0054 Boehringer Ingelheim Investigational Site, Harlingen, Texas
  - 1100.1486.0009 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1100.1486.0046 Boehringer Ingelheim Investigational Site, Annandale, Virginia
- Argentina (8):
  - 1100.1486.5401 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1486.5402 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1486.5404 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1486.5407 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1486.5408 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1486.5403 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1100.1486.5409 Boehringer Ingelheim Investigational Site, Quilmes
  - 1100.1486.5405 Boehringer Ingelheim Investigational Site, Rosario
- Australia (4):
  - 1100.1486.6101 Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - 1100.1486.6102 Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - 1100.1486.6104 Boehringer Ingelheim Investigational Site, Surry Hills, New South Wales
  - 1100.1486.6103 Boehringer Ingelheim Investigational Site, Brisbane, Queensland
- Belgium (9):
  - 1100.1486.3208 Boehringer Ingelheim Investigational Site, Bruges
  - 1100.1486.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1100.1486.3203 Boehringer Ingelheim Investigational Site, Brussels
  - 1100.1486.3205 Boehringer Ingelheim Investigational Site, Brussels
  - 1100.1486.3207 Boehringer Ingelheim Investigational Site, Brussels
  - 1100.1486.3209 Boehringer Ingelheim Investigational Site, Charleroi
  - 1100.1486.3202 Boehringer Ingelheim Investigational Site, Ghent
  - 1100.1486.3204 Boehringer Ingelheim Investigational Site, Liège
  - 1100.1486.3206 Boehringer Ingelheim Investigational Site, Liège
- Botswana (3):
  - 1100.1486.2605 Boehringer Ingelheim Investigational Site, Francistown
  - 1100.1486.2601 Boehringer Ingelheim Investigational Site, Gaborone
  - 1100.1486.2603 Boehringer Ingelheim Investigational Site, Gaborone
- Canada (8):
  - 1100.1486.1002 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1100.1486.1004 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1100.1486.1013 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1100.1486.1016 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1100.1486.1005 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1100.1486.1010 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1100.1486.1014 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1100.1486.1011 Boehringer Ingelheim Investigational Site, Quebec (Ste Foy), Quebec
- France (36):
  - 1100.1486.3305A Boehringer Ingelheim Investigational Site, Angers
  - 1100.1486.3305B Boehringer Ingelheim Investigational Site, Angers
  - 1100.1486.3307A Boehringer Ingelheim Investigational Site, Bondy
  - 1100.1486.3317A Boehringer Ingelheim Investigational Site, Bordeaux
  - 1100.1486.3316A Boehringer Ingelheim Investigational Site, Brest
  - 1100.1486.3316B Boehringer Ingelheim Investigational Site, Brest
  - 1100.1486.3314E Boehringer Ingelheim Investigational Site, Caen
  - 1100.1486.3304A Boehringer Ingelheim Investigational Site, Clamart
  - 1100.1486.3308A Boehringer Ingelheim Investigational Site, Lyon
  - 1100.1486.3308C Boehringer Ingelheim Investigational Site, Lyon
  - 1100.1486.3301A Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301B Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301C Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301D Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301E Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301F Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301G Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301H Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3301I Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1486.3306A Boehringer Ingelheim Investigational Site, Nice
  - 1100.1486.3303A Boehringer Ingelheim Investigational Site, Paris
  - 1100.1486.3303B Boehringer Ingelheim Investigational Site, Paris
  - 1100.1486.3303C Boehringer Ingelheim Investigational Site, Paris
  - 1100.1486.3303D Boehringer Ingelheim Investigational Site, Paris
  - 1100.1486.3312A Boehringer Ingelheim Investigational Site, Paris
  - 1100.1486.3312B Boehringer Ingelheim Investigational Site, Paris
  - 1100.1486.3309A Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1100.1486.3309B Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1100.1486.3318A Boehringer Ingelheim Investigational Site, Toulon
  - 1100.1486.3318B Boehringer Ingelheim Investigational Site, Toulon
  - 1100.1486.3318C Boehringer Ingelheim Investigational Site, Toulon
  - 1100.1486.3318D Boehringer Ingelheim Investigational Site, Toulon
  - 1100.1486.3302A Boehringer Ingelheim Investigational Site, Toulouse
  - 1100.1486.3302B Boehringer Ingelheim Investigational Site, Toulouse
  - 1100.1486.3302C Boehringer Ingelheim Investigational Site, Toulouse
  - 1100.1486.3310A Boehringer Ingelheim Investigational Site, Villeneuve-Saint-Georges
- Germany (29):
  - 1100.1486.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1486.4928 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1486.4932 Boehringer Ingelheim Investigational Site, Bochum
  - 1100.1486.4922 Boehringer Ingelheim Investigational Site, Bonn
  - 1100.1486.4907 Boehringer Ingelheim Investigational Site, Cologne
  - 1100.1486.4924 Boehringer Ingelheim Investigational Site, Cologne
  - 1100.1486.4911 Boehringer Ingelheim Investigational Site, Dortmund
  - 1100.1486.4919 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1100.1486.4908 Boehringer Ingelheim Investigational Site, Erlangen
  - 1100.1486.4906 Boehringer Ingelheim Investigational Site, Essen
  - 1100.1486.4926 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1100.1486.4916 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1100.1486.4929 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1100.1486.4901 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1100.1486.4930 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1100.1486.4909 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1486.4920 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1486.4925 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1486.4915 Boehringer Ingelheim Investigational Site, Hanover
  - 1100.1486.4923 Boehringer Ingelheim Investigational Site, Hanover
  - 1100.1486.4910 Boehringer Ingelheim Investigational Site, Kiel
  - 1100.1486.4927 Boehringer Ingelheim Investigational Site, Mainz
  - 1100.1486.4903 Boehringer Ingelheim Investigational Site, München
  - 1100.1486.4904 Boehringer Ingelheim Investigational Site, München
  - 1100.1486.4912 Boehringer Ingelheim Investigational Site, München
  - 1100.1486.4905 Boehringer Ingelheim Investigational Site, Münster
  - 1100.1486.4918 Boehringer Ingelheim Investigational Site, Osnabrück
  - 1100.1486.4913 Boehringer Ingelheim Investigational Site, Ulm/Donau
  - 1100.1486.4914 Boehringer Ingelheim Investigational Site, Würzburg
- Ireland (2):
  - 1100.1486.3531 Boehringer Ingelheim Investigational Site, Dublin
  - 1100.1486.3532 Boehringer Ingelheim Investigational Site, Dublin
- Italy (5):
  - 1100.1486.3908 Boehringer Ingelheim Investigational Site, Palermo
  - 1100.1486.3905 Boehringer Ingelheim Investigational Site, Pescara
  - 1100.1486.3901 Boehringer Ingelheim Investigational Site, Torino
  - 1100.1486.3907 Boehringer Ingelheim Investigational Site, Treviso
  - 1100.1486.3906 Boehringer Ingelheim Investigational Site, Verbania
- Mexico (2):
  - 1100.1486.5207 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1100.1486.5204 Boehringer Ingelheim Investigational Site, León
- Netherlands (4):
  - 1100.1486.3107 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1100.1486.3103 Boehringer Ingelheim Investigational Site, Arnhem
  - 1100.1486.3101 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1100.1486.3102 Boehringer Ingelheim Investigational Site, Zwolle
- Poland (3):
  - 1100.1486.4803 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1100.1486.4801 Boehringer Ingelheim Investigational Site, Chorzów
  - 1100.1486.4804 Boehringer Ingelheim Investigational Site, Warsaw
- Portugal (3):
  - 1100.1486.3503 Boehringer Ingelheim Investigational Site, Amadora
  - 1100.1486.3501 Boehringer Ingelheim Investigational Site, Lisbon
  - 1100.1486.3504 Boehringer Ingelheim Investigational Site, Lisbon
- Puerto Rico (2):
  - 1100.1486.0024 Boehringer Ingelheim Investigational Site, Ponce
  - 1100.1486.0033 Boehringer Ingelheim Investigational Site, San Juan
- Romania (2):
  - 1100.1486.4001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1100.1486.4002 Boehringer Ingelheim Investigational Site, Bucharest
- Russia (2):
  - 1100.1486.7002 Boehringer Ingelheim Investigational Site, Moscow
  - 1100.1486.7001 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Africa (10):
  - 1100.1486.2707 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 1100.1486.2712 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 1100.1486.2703 Boehringer Ingelheim Investigational Site, Cape Town
  - 1100.1486.2709 Boehringer Ingelheim Investigational Site, Cape Town
  - 1100.1486.2711 Boehringer Ingelheim Investigational Site, Cape Town
  - 1100.1486.2701 Boehringer Ingelheim Investigational Site, Edenvale
  - 1100.1486.2710 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1100.1486.2706 Boehringer Ingelheim Investigational Site, Mbombela
  - 1100.1486.2702 Boehringer Ingelheim Investigational Site, Port Elizabeth
  - 1100.1486.2704 Boehringer Ingelheim Investigational Site, Pretoria
- Spain (13):
  - 1100.1486.3406 Boehringer Ingelheim Investigational Site, Alcalá de Henares (Madrid)
  - 1100.1486.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1486.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1486.3410 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1486.3415 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1486.3417 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1486.3404 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1100.1486.3403 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1486.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1486.3407 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1486.3414 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1486.3416 Boehringer Ingelheim Investigational Site, Mataró
  - 1100.1486.3408 Boehringer Ingelheim Investigational Site, Valencia
- Switzerland (8):
  - 1100.1486.4101 Boehringer Ingelheim Investigational Site, Basel
  - 1100.1486.4109 Boehringer Ingelheim Investigational Site, Bern
  - 1100.1486.4107 Boehringer Ingelheim Investigational Site, Geneva
  - 1100.1486.4106 Boehringer Ingelheim Investigational Site, La Chaux-de-Fonds
  - 1100.1486.4104 Boehringer Ingelheim Investigational Site, Lausanne
  - 1100.1486.4102 Boehringer Ingelheim Investigational Site, Lugano
  - 1100.1486.4108 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 1100.1486.4110 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (8):
  - 1100.1486.4406 Boehringer Ingelheim Investigational Site, Birmingham
  - 1100.1486.4403 Boehringer Ingelheim Investigational Site, London
  - 1100.1486.4404 Boehringer Ingelheim Investigational Site, London
  - 1100.1486.4405 Boehringer Ingelheim Investigational Site, London
  - 1100.1486.4407 Boehringer Ingelheim Investigational Site, London
  - 1100.1486.4401 Boehringer Ingelheim Investigational Site, Manchester
  - 1100.1486.4408 Boehringer Ingelheim Investigational Site, Manchester
  - 1100.1486.4402 Boehringer Ingelheim Investigational Site, Plaistow, London

REFERENCES:
- [Derived] Gathe J, Andrade-Villanueva J, Santiago S, Horban A, Nelson M, Cahn P, Bogner J, Spencer D, Podzamczer D, Yong CL, Nguyen T, Zhang W, Drulak M, Quinson AM. Efficacy and safety of nevirapine extended-release once daily versus nevirapine immediate-release twice-daily in treatment-naive HIV-1-infected patients. Antivir Ther. 2011;16(5):759-69. doi: 10.3851/IMP1803. PMID 21817198

RESULTS

PARTICIPANT FLOW:
Groups:
- NVP IR 200mg QD: Nevirapine immediate release 200 mg given once daily
- NVP IR 200mg BID: Nevirapine immediate release 200 mg given twice daily
- NVP XR 400mg QD: Nevirapine extended release 400 mg given once daily
Period: 14 Day Lead-In Period
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD | NVP XR | NVP IR to XR
Started | 1068 | 0 | 0 | 0 | 0
Completed | 1013 | 0 | 0 | 0 | 0
Not Completed | 55 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 38 | 0 | 0 | 0 | 0
Not completed — In/Exclusion criteria | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 0 | 0 | 0 | 0
Period: 144-week Double-blind, Double-dummy
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD | NVP XR | NVP IR to XR
Started | 0 | 508 | 505 | 0 | 0
Completed | 0 | 358 | 378 | 0 | 0
Not Completed | 0 | 150 | 127 | 0 | 0
Not completed — Adverse Event | 0 | 48 | 43 | 0 | 0
Not completed — Protocol Violation | 0 | 15 | 9 | 0 | 0
Not completed — Lost to Follow-up | 0 | 15 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 19 | 7 | 0 | 0
Not completed — Lack of Efficacy | 0 | 36 | 33 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 9 | 0 | 0
Not completed — Death | 0 | 6 | 3 | 0 | 0
Not completed — Not treated with study drug | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 8 | 11 | 0 | 0
Period: Open-Label Extension Period
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD | NVP XR | NVP IR to XR
Started | 0 | 1 | 0 | 358 | 378
Completed | 0 | 1 | 0 | 315 | 328
Not Completed | 0 | 0 | 0 | 43 | 50
Not completed — Declined entry into extension period | 0 | 0 | 0 | 43 | 50

BASELINE CHARACTERISTICS:
Groups:
- NVP IR 200mg QD: Nevirapine immediate release 200 mg tablets given once daily
- NVP IR 200mg BID: Nevirapine immediate release 200 mg tablets given twice daily
- NVP XR 400mg QD: Nevirapine extended release 400 mg tablets given once daily
- Total: Total of all reporting groups
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD | Total
Number analyzed (Participants) | 0 | 508 | 505 | 1013
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 38.0 (9.7) | 38.3 (9.7) | 38.1 (9.7)
Age, Customized [Number; unit: participants]
  18 to < 41 years |  | 316 | 299 | 615
  41 to < 56 years |  | 165 | 182 | 347
  56 to < 65 years |  | 25 | 19 | 44
  65 years or more |  | 2 | 5 | 7
Gender [Number; unit: participants]
  Female |  | 75 | 74 | 149
  Male |  | 433 | 431 | 864
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaskan Native |  | 6 | 8 | 14
  Asian |  | 13 | 15 | 28
  Black |  | 113 | 94 | 207
  Hawaiian / Pacific Isle. |  | 0 | 1 | 1
  White |  | 376 | 387 | 763
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic / Latino |  | 109 | 115 | 224
  Not Hispanic / Latino |  | 399 | 390 | 789
Region of Enrollment [Number; unit: participants]
  North America / Australia |  | 149 | 141 | 290
  Europe |  | 253 | 257 | 510
  Latin America |  | 49 | 58 | 107
  Africa |  | 57 | 49 | 106
Smoking History [Number; unit: participants]
  Never smoked |  | 250 | 224 | 474
  Ex-smoker |  | 81 | 86 | 167
  Current smoker |  | 177 | 195 | 372
Alcohol Status [Number; unit: participants]
  Non drinker |  | 151 | 168 | 319
  Drinks - no interfere with trial |  | 354 | 335 | 689
  Drinks - could interfere with trial |  | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Proportion of Virologic Response at Week 48 Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Primary endpoint was the number of patients with a sustained virologic response through week 48 using LLOQ = 50 copies/mL
Time Frame: week 48
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of blinded medication
Measure: Number; unit: participants
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD
Number analyzed (Participants) | 0 | 506 | 505
participants
  Responder |  | 384 | 409
  Non responder |  | 122 | 96
Statistical Analysis 1: Comparison: NVP IR 200mg BID vs NVP XR 400mg QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of nevirapine XR to nevirapine IR was established if the lower bound of the confidence interval was greater than -10%; p < 0.0001, Cochran's statistic; Cochran's statistic = 4.9, 95% CI [-0.1 to 10.0] — Weighted treatment difference and corresponding variance were calculated based on Cochran's statistic

2. Secondary Outcome: Kaplan-Meier Estimates of the Proportions of Patients Without Loss of Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Time Frame: week 0 to 144
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD
Number analyzed (Participants) | 0 | 506 | 505
proportion of participants
  Interval Week 0 to <2 |  | 1 | 1
  Interval Week 2 to <4 |  | 0.84 | 0.865
  Interval Week 4 to <6 |  | 0.838 | 0.865
  Interval Week 6 to <8 |  | 0.834 | 0.865
  Interval Week 8 to <12 |  | 0.834 | 0.863
  Interval Week 12 to <16 |  | 0.832 | 0.861
  Interval Week 16 to <24 |  | 0.83 | 0.859
  Interval Week 24 to <32 |  | 0.822 | 0.848
  Interval Week 32 to <40 |  | 0.806 | 0.832
  Interval Week 40 to <48 |  | 0.792 | 0.816
  Interval Week 48 to <60 |  | 0.777 | 0.808
  Interval Week 60 to <72 |  | 0.759 | 0.788
  Interval Week 72 to <84 |  | 0.733 | 0.766
  Interval Week 84 to <96 |  | 0.713 | 0.745
  Interval Week 96 to <108 |  | 0.686 | 0.719
  Interval Week 108 to <120 |  | 0.662 | 0.697
  Interval Week 120 to <132 |  | 0.65 | 0.681
  Interval Week 132 to <144 |  | 0.63 | 0.671
  Interval Week 144 to <168 |  | 0.61 | 0.66

3. Secondary Outcome: Proportion of Sustained Virologic Response at Week 144 Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 144 using LLOQ = 50 copies/mL
Time Frame: week 144
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD
Number analyzed (Participants) | 0 | 506 | 505
participants
  Responder |  | 296 | 321
  Non responder |  | 210 | 184
Statistical Analysis 1: Comparison: NVP IR 200mg BID vs NVP XR 400mg QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of nevirapine XR to nevirapine IR was established if the lower bound of the confidence interval was greater than -2%; p < 0.0001, Cochran's statistic; Cochran's statistic = 4.84, 95% CI [-1.11 to 10.79] — Weighted treatment difference and corresponding variance were calculated based on Cochran's statistic

4. Secondary Outcome: Kaplan-Meier Estimates for Time to New AIDS or AIDS-related Progression Event or Death, Full Analysis Set Population
Time Frame: week 0 to 144
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD
Number analyzed (Participants) | 0 | 506 | 505
proportion of participants
  Interval Week 0 to <2 |  | 0 | 0
  Interval Week 2 to <4 |  | 0.006 | 0.002
  Interval Week 4 to <6 |  | 0.006 | 0.006
  Interval Week 6 to <8 |  | 0.023 | 0.008
  Interval Week 8 to <12 |  | 0.029 | 0.01
  Interval Week 12 to <16 |  | 0.029 | 0.019
  Interval Week 16 to <24 |  | 0.031 | 0.021
  Interval Week 24 to <32 |  | 0.04 | 0.025
  Interval Week 32 to <40 |  | 0.042 | 0.025
  Interval Week 40 to <48 |  | 0.047 | 0.027
  Interval Week 48 to <60 |  | 0.047 | 0.027
  Interval Week 60 to <72 |  | 0.052 | 0.032
  Interval Week 72 to <84 |  | 0.054 | 0.035
  Interval Week 84 to <96 |  | 0.054 | 0.04
  Interval Week 96 to <108 |  | 0.057 | 0.04
  Interval Week 108 to <120 |  | 0.057 | 0.045
  Interval Week 120 to <132 |  | 0.06 | 0.047
  Interval Week 132 to <144 |  | 0.06 | 0.047
  Interval Week 144 to <168 |  | 0.062 | 0.047

5. Secondary Outcome: Comparison of HIV-1 Viral Load (log10 Copies/mL) Change From Baseline at Week 144, Full Analysis Set Population
Time Frame: baseline, week 144
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of blinded medication; descriptive analysis uses the imputation method: last observation carried forward; statistical analysis uses observed cases
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD
Number analyzed (Participants) | 0 | 506 | 505
log10 copies/mL |  | -2.7 (0.9) | -2.8 (0.8)
Statistical Analysis 1: Comparison: NVP IR 200mg BID vs NVP XR 400mg QD; Test type: Superiority or Other; p = 0.7719, ANCOVA; Means adjusted for baseline HIV-1 viral load stratum; Mean Difference (Final Values) = -0.01, 95% CI [-0.08 to 0.06]

6. Secondary Outcome: Comparison of CD4+ Cell Count (Cells/Cubic Millimeter) Change From Baseline at Week 144, Full Analysis Set Population
Time Frame: baseline, week 144
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | NVP IR 200mg QD | NVP IR 200mg BID | NVP XR 400mg QD
Number analyzed (Participants) | 0 | 506 | 505
cells/cubic millimeter |  | 239.3 (171.4) | 270.7 (183.1)
Statistical Analysis 1: Comparison: NVP IR 200mg BID vs NVP XR 400mg QD; Test type: Superiority or Other; p = 0.0078, ANCOVA; Means adjusted for baseline HIV-1 viral load stratum; Mean Difference (Final Values) = 32.87, 95% CI [8.67 to 57.06]

7. Secondary Outcome: Occurrence of Rashes
Description: Frequency of patients with drug related rash events by functional grouping
Time Frame: until last patient completed 144 weeks (up to 193 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- NVP IR: Patients received nevirapine IR during the 144 week blinded phase and nevirapine XR during open label extension
- NVP XR: Patients receiving nevirapine XR during the 144 week blinded phase and nevirapine XR during open label extension
- IR-IR/XR: Patients receiving nevirapine IR during the 144 week blinded phase and then receiving nevirapine XR in the post week 144 of extension
- XR-IR/XR: Patients receiving nevirapine XR during open label extension and previously receiving nevirapine IR during the pre week 144
Arm/Group | NVP IR | NVP XR | IR-IR/XR | XR-IR/XR
Number analyzed (Participants) | 191 | 505 | 315 | 315
participants
  rash group I | 9 | 11 | 6 | 0
  rash group II | 6 | 13 | 3 | 0
  rash group IIA | 4 | 5 | 1 | 0
  rash group III | 3 | 5 | 0 | 0
  rash group IV | 0 | 0 | 0 | 0

8. Secondary Outcome: Occurrence of Elevations in Laboratory Measurement by DAIDS Grade
Time Frame: until last patient completed 144 weeks (up to 193 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NVP IR | NVP XR | IR-IR/XR | XR-IR/XR
Number analyzed (Participants) | 191 | 505 | 315 | 315
participants
  DAIDS grade 3 or 4 AEs | 53 | 111 | 71 | 8
  DAIDS grade 4 AEs | 17 | 25 | 11 | 3

9. Secondary Outcome: Kaplan -Meier Estimate of Cumulative Probability of Permanent Discontinuation of Study Medication
Time Frame: week 0 to 144
Population: as for outcome 1
Measure: Number; unit: cumulative probability
Groups:
- NVP IR: Nevirapine immediate release 200 mg tablets given twice daily
- NVP XR: Nevirapine extended release 400 mg tablets given once daily
Arm/Group | NVP IR | NVP XR
Number analyzed (Participants) | 506 | 505
cumulative probability
  Interval Week 0 to <2 | 0.000 | 0.000
  Interval Week 2 to <4 | 0.000 | 0.000
  Interval Week 4 to <6 | 0.034 | 0.026
  Interval Week 6 to <8 | 0.067 | 0.046
  Interval Week 8 to <12 | 0.081 | 0.059
  Interval Week 12 to <16 | 0.093 | 0.067
  Interval Week 16 to <24 | 0.113 | 0.083
  Interval Week 24 to <32 | 0.130 | 0.115
  Interval Week 32 to <40 | 0.156 | 0.139
  Interval Week 40 to <48 | 0.172 | 0.156
  Interval Week 48 to <60 | 0.192 | 0.162
  Interval Week 60 to <72 | 0.202 | 0.176
  Interval Week 72 to <84 | 0.213 | 0.188
  Interval Week 84 to <96 | 0.229 | 0.206
  Interval Week 96 to <108 | 0.243 | 0.218
  Interval Week 108 to <120 | 0.267 | 0.232
  Interval Week 120 to <132 | 0.275 | 0.236
  Interval Week 132 to <144 | 0.289 | 0.244

10. Secondary Outcome: Kaplan -Meier Estimate of Cumulative Probability of Grade 3 or 4 ALT/AST Abnormalities
Time Frame: week 0 to 72
Population: Treated set (TS) includes all patients who were dispensed study medication and were documented to have taken at least one doe of investigational treatment, including the lead in nevirapine dose
Measure: Number; unit: cumulative probability
Arm/Group | NVP IR | NVP XR
Number analyzed (Participants) | 506 | 505
cumulative probability
  Interval Week 0 to <2 | 0.000 | 0.000
  Interval Week 2 to <4 | 0.000 | 0.002
  Interval Week 4 to <6 | 0.012 | 0.014
  Interval Week 6 to <8 | 0.049 | 0.026
  Interval Week 8 to <12 | 0.059 | 0.034
  Interval Week 12 to <16 | 0.063 | 0.036
  Interval Week 16 to <24 | 0.063 | 0.036
  Interval Week 24 to <32 | 0.067 | 0.043
  Interval Week 32 to <40 | 0.070 | 0.049
  Interval Week 40 to <48 | 0.076 | 0.056
  Interval Week 48 to <60 | 0.076 | 0.058
  Interval Week 60 to <72 | 0.076 | 0.058
  Interval Week >=72 | 0.076 | 0.070

11. Secondary Outcome: Kaplan -Meier Estimate of Cumulative Probability of Grade 3 or 4 Asymptotic Transaminases Abnormalities
Time Frame: week 0 to 72
Population: as for outcome 10
Measure: Number; unit: cumulative probability
Arm/Group | NVP IR | NVP XR
Number analyzed (Participants) | 506 | 505
cumulative probability
  Interval Week 0 to <2 | 0.000 | 0.000
  Interval Week 2 to <4 | 0.000 | 0.000
  Interval Week 4 to <6 | 0.006 | 0.002
  Interval Week 6 to <8 | 0.027 | 0.006
  Interval Week 8 to <12 | 0.033 | 0.008
  Interval Week 12 to <16 | 0.039 | 0.008
  Interval Week 16 to <24 | 0.039 | 0.008
  Interval Week 24 to <32 | 0.042 | 0.015
  Interval Week 32 to <40 | 0.044 | 0.019
  Interval Week 40 to <48 | 0.053 | 0.028
  Interval Week 48 to <60 | 0.053 | 0.031
  Interval Week 60 to <72 | 0.053 | 0.033
  Interval Week >=72 | 0.053 | 0.033

12. Secondary Outcome: Kaplan -Meier Estimate of Cumulative Probability of Clinical Hepatic Events
Time Frame: week 0 to 72
Population: as for outcome 10
Measure: Number; unit: cumulative probability
Arm/Group | NVP IR | NVP XR
Number analyzed (Participants) | 506 | 505
cumulative probability
  Interval Week 0 to <2 | 0.000 | 0.000
  Interval Week 2 to <4 | 0.000 | 0.002
  Interval Week 4 to <6 | 0.012 | 0.010
  Interval Week 6 to <8 | 0.022 | 0.016
  Interval Week 8 to <12 | 0.024 | 0.018
  Interval Week 12 to <16 | 0.026 | 0.018
  Interval Week 16 to <24 | 0.026 | 0.018
  Interval Week 24 to <32 | 0.026 | 0.020
  Interval Week 32 to <40 | 0.026 | 0.022
  Interval Week 40 to <48 | 0.029 | 0.022
  Interval Week 48 to <60 | 0.029 | 0.022
  Interval Week 60 to <72 | 0.032 | 0.022
  Interval Week >=72 | 0.038 | 0.026

13. Secondary Outcome: Kaplan -Meier Estimate of Cumulative Probability of Group III or IV Drug-related Rash
Time Frame: week 0 to 72
Population: as for outcome 10
Measure: Number; unit: cumulative probability
Arm/Group | NVP IR | NVP XR
Number analyzed (Participants) | 506 | 505
cumulative probability
  Interval Week 0 to <2 | 0.000 | 0.000
  Interval Week 2 to <4 | 0.000 | 0.000
  Interval Week 4 to <6 | 0.002 | 0.006
  Interval Week 6 to <8 | 0.004 | 0.008
  Interval Week 8 to <12 | 0.004 | 0.010
  Interval Week 12 to <16 | 0.004 | 0.010
  Interval Week 16 to <24 | 0.004 | 0.010
  Interval Week 24 to <32 | 0.004 | 0.010
  Interval Week 32 to <40 | 0.004 | 0.010
  Interval Week 40 to <48 | 0.004 | 0.010
  Interval Week 48 to <60 | 0.004 | 0.010
  Interval Week 60 to <72 | 0.004 | 0.010
  Interval Week >=72 | 0.004 | 0.010

14. Secondary Outcome: Relative Bioavailability Trough C_pre,ss,1
Description: Relative bioavailability measured of trough concentrations. Analysis based on adjusted by-treatment geometric means, the adjusted geometric mean ratio of NVP XR : NVP IR and it's 90% confidence interval with p-value and the inter-individual geometric coefficient of variation.
Time Frame: week 132
Population: Only patients with trough drawn PK time window (12+/-2.5 hr for IR; 24+/-5hr for XR) at week 132 are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | NVP IR | NVP XR
Number analyzed (Participants) | 276 | 311
ng/mL | 4567.03 (49.9) | 3634.26 (49.9)
Statistical Analysis 1: Comparison: NVP IR vs NVP XR; adjusted geometric mean ratio NVP XR : NVP IR; Test type: Non-Inferiority or Equivalence — equivalence test with 80% -125% boundaries; p = 0.5542, ANOVA — p-value for ratio outside the interval 80%-125%; adjusted gMean = 79.58, 90% CI [74.62 to 84.86], Standard Error of Mean 1.04 — Inter-individual gCV = 49.9

15. Secondary Outcome: Occurrence of Hepatic Events
Description: Frequency of patients with hepatitis symptoms
Time Frame: until last patient completed 144 weeks (up to 193 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- NVP IR: Patients received nevirapine IR during the 144 week blinded phase but who never took nevirapine XR during the open label extension
- XR-IR/XR: Patients receiving nevirapine XR during open label extension who had previously received nevirapine IR during the pre week 144
Arm/Group | NVP IR | NVP XR | IR-IR/XR | XR-IR/XR
Number analyzed (Participants) | 191 | 505 | 315 | 315
participants | 10 | 8 | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 193 weeks
Description: Safety data in this report included all the patient visits up to the point in time when the last patient completed 144 weeks in the trial. This also includes safety data for patient visits in the post week 144 open label extension which patients in either treatment group who completed the 144 week blinded phase could enter (see also Limitation).
Groups:
- NVP IR-IR/XR: Patients receiving nevirapine IR during the 144 week blinded phase and then receiving nevirapine XR in the post week 144 of extension
- NVP XR-IR/XR: Patients receiving nevirapine XR during open label extension who had previously receiving nevirapine IR during the pre week 144
Arm/Group | NVP IR 200mg QD | NVP IR | NVP XR | NVP IR-IR/XR | NVP XR-IR/XR
Serious Adverse Events (participants affected / at risk) | 20/1068 | 33/191 | 93/505 | 50/315 | 9/315
Other Adverse Events (participants affected / at risk) | 308/1068 | 131/191 | 403/505 | 271/315 | 81/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVP IR 200mg QD (N=1068) | NVP IR (N=191) | NVP XR (N=505) | NVP IR-IR/XR (N=315) | NVP XR-IR/XR (N=315)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial rub (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 1 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 1 | 0
Hyperplasia (General disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Polyserositis (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 2 | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
AIDS encephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Eye infection syphilitic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningitis histoplasma (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Neurocryptococcosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 7 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 3 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Syphilis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Catheterisation cardiac normal (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Epithelioid sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Osteosarcoma localised (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervical root pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intracranial hypotension (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 4 | 3 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Social phobia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Infertility female (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0 | 0
Aborted pregnancy (Social circumstances) | 0 | 0 | 0 | 1 | 0
Alcohol use (Social circumstances) | 0 | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 2 | 1 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Removal of internal fixation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Secondary hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVP IR 200mg QD (N=1068) | NVP IR (N=191) | NVP XR (N=505) | NVP IR-IR/XR (N=315) | NVP XR-IR/XR (N=315)
Abdominal pain (Gastrointestinal disorders) | 8 | 7 | 25 | 25 | 2
Diarrhoea (Gastrointestinal disorders) | 27 | 27 | 94 | 63 | 7
Nausea (Gastrointestinal disorders) | 71 | 18 | 38 | 38 | 3
Vomiting (Gastrointestinal disorders) | 16 | 11 | 35 | 22 | 1
Fatigue (General disorders) | 40 | 10 | 34 | 28 | 2
Pyrexia (General disorders) | 20 | 12 | 25 | 12 | 2
Bronchitis (Infections and infestations) | 7 | 12 | 71 | 35 | 4
Gastroenteritis (Infections and infestations) | 5 | 10 | 36 | 27 | 2
Herpes zoster (Infections and infestations) | 6 | 7 | 26 | 17 | 1
Influenza (Infections and infestations) | 5 | 9 | 33 | 25 | 0
Nasopharyngitis (Infections and infestations) | 10 | 17 | 123 | 87 | 15
Pharyngitis (Infections and infestations) | 5 | 7 | 33 | 23 | 2
Sinusitis (Infections and infestations) | 5 | 5 | 37 | 22 | 2
Syphilis (Infections and infestations) | 1 | 8 | 28 | 19 | 7
Upper respiratory tract infection (Infections and infestations) | 13 | 23 | 83 | 50 | 12
Urinary tract infection (Infections and infestations) | 2 | 4 | 26 | 12 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 33 | 25 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 40 | 30 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 16 | 20 | 2
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 29 | 16 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 19 | 16 | 1
Headache (Nervous system disorders) | 58 | 18 | 61 | 55 | 3
Anxiety (Psychiatric disorders) | 5 | 7 | 20 | 16 | 2
Depression (Psychiatric disorders) | 8 | 7 | 37 | 31 | 6
Insomnia (Psychiatric disorders) | 8 | 9 | 27 | 19 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 52 | 36 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 30 | 13 | 3
Rash (Skin and subcutaneous tissue disorders) | 74 | 26 | 56 | 25 | 2
Hypertension (Vascular disorders) | 5 | 13 | 38 | 22 | 3

LIMITATIONS AND CAVEATS:
For the lead-in-period with NVP IR 200mg QD, MedDRA Version 12.1 was used for AE/SAE reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.